CLINICAL TRIAL: NCT01830283
Title: Phase 4 Study of the Varicella Vaccine After the 2nd Dose Vaccination
Brief Title: The Safety, Immunogenicity and Immune Effect Research of the Varicella Vaccine After the 2nd Dose Vaccination
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beijing Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BJCDPC-8
Record Dates: First submitted 2013-04-03; First posted 2013-04-12 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-04

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox | interventions — Chickenpox Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 dose varicella vaccine (Active Comparator): The providers would get the 2nd dose since they had one dose varicella vaccine
  Interventions: Biological: varicella vaccine
- 2 dose varicella vaccine (Experimental): The provider never get the varicella vaccine
  Interventions: Biological: varicella vaccine

INTERVENTIONS:
Biological: varicella vaccine — The providers would get varicella vaccine

SUMMARY:
To investigate the safety, immunogenicity and immune effect of the Varicella vaccine after the 2nd dose vaccination in Chao yang district, Bei jing, since the 2nd varicella vaccination was promoted by Beijing Center for Disease Control and Prevention in November, 2012.

DETAILED DESCRIPTION:
"Breakthrough" varicella cases and varicella cases were monitored to evaluate the protective effective in a large population.

Make the basic evaluation of safety for the two dose of varicella vaccination

Monitoring the Varicella virus origin and virus types from illness cases in Chao yang district

Make the evaluation of healthy costs reduce for the varicella emergency vaccination after large number of varicella cases occurred.

ELIGIBILITY:
Inclusion Criteria:

* Participants were between 4-12 years old
* Participants were in good healthy determined through medical history, physical examination, clinical judgment of the investor

Exclusion Criteria:

* Having a fever (axillary temperature >37.0℃) before enrollment;
* Having a disease history of seizures, brain and mental disease and the vaccination history of allergies and convulsions;
* Antibiotics allergy;
* Having a problem of intramuscular injection because thrombocytopenia or other blood coagulation disorder;
* Having immunodeficiency or under immunosuppression therapy, radiation therapy;
* Having respiratory diseases, acute infection, chronic disease and HIV infection;
* Having systemic skin rash, skin tinea, herpes;
* Chronic liver and kidney disease;
* Heart disease, and severe hypertension;
* Have received whole blood, plasma or immunoglobulin therapy 3 months before enrollment;
* Have not received other vaccination in 7 days before enrollment

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50000 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-06 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of varicella after 2 dose vaccination | 5 years
  Detection the Varicella virus origin and virus types from illness cases in Chao yang district

SECONDARY OUTCOMES:
Adverse event rate of varicella vaccine after 2 dose injection | 5 years
  Adverse event rate of varicella vaccine after 2 dose injection

OTHER OUTCOMES:
Antibody titre of varicella vaccine after 2 dose injection | 6 monthes
  Antibody titre of varicella vaccine after 2 dose injection

CONTACTS AND LOCATIONS:
Overall Officials: Nianmin Shi, Principal Investigator — Beijing Chaoyang District Centers for Disease Control and Prevention
Locations (1):
- Beijing Chaoyang District Centers for Disease Control and Prevention, Beijing, China